CLINICAL TRIAL: NCT02354248
Title: Application of the Triple Stimulation Technique to Patients With CNS Disorders Including Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Bernard Dachy, Head of clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-TST01
Record Dates: First submitted 2015-01-23; First posted 2015-02-03 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Stroke Patients
Keywords: TST; TMS; Stroke patients; EMG

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke patients (Experimental): The patients will be submitted to a triple stimulation examination.
  Interventions: Procedure: Triple stimulation technique
- Control Subjects (Active Comparator): This group of patients did not suffer from a stroke. They will also be submitted to a triple stimulation examination.
  Interventions: Procedure: Triple stimulation technique

INTERVENTIONS:
Procedure: Triple stimulation technique — Evoked motor potentials obtained by magnetic transcranial stimulation are usually used, in standard practice, to evaluate the corticospinal tract. This procedure combines two techniques: the magnetic stimulation and the electroneuromyography. It is based on the double collision principle between the descending central stimulation (magnetic) and the ascending peripheric stimulation, hereby suppressing the issue of desynchronisation of evoked motor potentials. The Triple stimulation technique allows a better quantification of the proportion of motor units activated by the transcranial stimulation.

SUMMARY:
TST (Triple stimulation technique) helps to better quantify the proportion of motor units activated by transcranial magnetic stimulation. The abnormal amplitude registered by TST is proportional to the intensity of conduction disorders. The evaluation of these disorders is more precise with this technique than with the slowing of the central conduction time (CCT).

The investigators propose to use this technique in CNS pathologies where this disorder is significant and essential, like multiple sclerosis and stroke.

ELIGIBILITY:
Inclusion Criteria:

* stroke patients with hemiparesia

Exclusion Criteria:

* pace maker
* epilepsia
* metallic neurosurgical implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

PRIMARY OUTCOMES:
Amplitude of the motor evoked potentials | during the TST (30 min)
Surface of the motor evoked potentials | during the TST (30 min)
Amplitude ratio of the TST | during the TST (30 min)
Surface ratio of the TST | during the TST (30 min)
TMS threshold | during TST (30 min)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Dachy, MD, Principal Investigator — CHU Brugmann; Andrey Bragin, MD, Principal Investigator — CHU Brugmann; Pedro Calderon, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Magistris MR, Rosler KM, Truffert A, Myers JP. Transcranial stimulation excites virtually all motor neurons supplying the target muscle. A demonstration and a method improving the study of motor evoked potentials. Brain. 1998 Mar;121 ( Pt 3):437-50. doi: 10.1093/brain/121.3.437. PMID 9549520
- [Background] Magistris MR, Rosler KM, Truffert A, Landis T, Hess CW. A clinical study of motor evoked potentials using a triple stimulation technique. Brain. 1999 Feb;122 ( Pt 2):265-79. doi: 10.1093/brain/122.2.265. PMID 10071055